CLINICAL TRIAL: NCT02056860
Title: Feasibility and Optimization of High Frequency Oscillation (HFO) for Detection of Lung Infections
Brief Title: Detecting Lung Infections Through Vibration
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 821-2013
Record Dates: First submitted 2014-01-30; First posted 2014-02-06 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Lung Infection
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group 1 will receive 15 Hz: Group 1 (n=30), these subjects will receive 10 minutes of High Frequency Oscillation at 15 Hz at .75 cm on day 1. Then will have a 24 hour washout. On day 2 will receive 10 minutes of low Frequency Oscillation at 15 Hz at 1.25 cm.
  Interventions: Procedure: Group 1 will receive 15 Hz
- Group 2 will receive 30 Hz: Group 2 (n=30), these subjects will receive 10 minutes of High Frequency Oscillation at 30 Hz at .75 cm on day 1. Then will have a 24 hour washout. On day 2 will receive 10 minutes of low Frequency Oscillation at 30 Hz 1.25 cm.
  Interventions: Procedure: Group 2 will receive 30 Hz
- Group 3 will receive 60 Hz: Group 3 (n=30), these subjects will receive 10 minutes of High Frequency Oscillation at 60 Hz 2 .75 cm on day 1. Then will have a 24 hour washout. On day 2 will receive 10 minutes of low Frequency Oscillation at 60 Hz at 1.25 cm.
  Interventions: Procedure: Group 3 will receive 60 Hz
- Group 4 will receive 100 Hz: Group 4 (n=30), these subjects will receive 10 minutes of High Frequency Oscillation at 100 Hz at .75 cm on day 1. Then will have a 24 hour washout. On day 2 will receive 10 minutes of low Frequency Oscillation at 100 Hz at 1.25 cm.
  Interventions: Procedure: Group 4 will receive 100 Hz
- Phase II Optimal Frequency: Participants in Phase II will undergo 10 minutes of HFO at the optimal frequency as determined during Phase I.
  Interventions: Procedure: Phase II Optimal Frequency

INTERVENTIONS:
Procedure: Group 1 will receive 15 Hz — Group 1 (n=30), these subjects will receive 10 minutes of High Frequency Oscillation at 15 Hz at .75 cm on day 1. Then will have a 24 hour washout. On day 2 will receive 10 minutes of low Frequency Oscillation at 15 Hz at 1.25 cm.
  Groups: Group 1 will receive 15 Hz
Procedure: Group 2 will receive 30 Hz — Group 2 (n=30), these subjects will receive 10 minutes of High Frequency Oscillation at 30 Hz at .75 cm on day 1. Then will have a 24 hour washout. On day 2 will receive 10 minutes of low Frequency Oscillation at 30 Hz 1.25 cm.
  Groups: Group 2 will receive 30 Hz
Procedure: Group 3 will receive 60 Hz — Group 3 (n=30), these subjects will receive 10 minutes of High Frequency Oscillation at 60 Hz .75 cm on day 1. Then will have a 24 hour washout. On day 2 will receive 10 minutes of low Frequency Oscillation at 60 Hz at 1.25 cm.
  Groups: Group 3 will receive 60 Hz
Procedure: Group 4 will receive 100 Hz — Group 4 (n=30), these subjects will receive 10 minutes of High Frequency Oscillation at 100 Hz at .75 cm on day 1. Then will have a 24 hour washout. On day 2 will receive 10 minutes of low Frequency Oscillation at 100 Hz at 1.25 cm.
  Groups: Group 4 will receive 100 Hz
Procedure: Phase II Optimal Frequency — Participants in Phase II will undergo 10 minutes of HFO at the optimal frequency as determined during Phase I.
  Groups: Phase II Optimal Frequency

SUMMARY:
The purpose of this study is to test a lung air vibrator device for vibrating air inside the lung. This exploratory diagnostic trial will test a novel and non-invasive means of detecting lower airway infections using exhaled breath sample.

DETAILED DESCRIPTION:
This study has two phases. Once the subject has consented phase 1 will start by the subject breathing air out of their lungs into the device. Next, the subject will simply breathe through the mouthpiece with the machine turned on and take samples of exhaled air.

In phase 2, the subjects will breathe air out of their lungs into the device for 15 minutes. Next, the subject will simply breathe through the mouthpiece with the machine turned on and take samples of exhaled air for 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50

Exclusion Criteria:

* History of major respiratory compromise (except cystic fibrosis if included within cystic fibrosis cohort)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy normal adults age 18 to 50 Individuals with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Optimal Operating Conditions for HFO Device | 6 months
  Following informed consent procedures, participants will be randomly assigned (much like a flip of a coin) to one of four experimental groups in order to test the effects of various frequencies of HFO on the size and concentration of particles obtained from EB. Group 1 (n=30) will receive 10 minutes of HFO at 15 Hz. Group 2 (n=30) will receive an identical course of HFO with the frequency set at 30 Hz. Group 3 (n=30) will receive HFO at 60 Hz and Group 4 (n=30) at 100 Hz. Participants will be tested on two separate days in order to systematically vary HFO intensity. Once again, much like a flip of a coin, each participant will be randomly assigned to receive HFO at either a low (0.75 cmH2O) or high (1.25 cm H2O) intensity on HFO Day 1. Participants receiving low intensity HFO on Day 1 will receive high intensity HFO on Day 2, and vice versa. Between HFO Testing Day 1 and 2 there will be a washout period of at least 24 hours.

SECONDARY OUTCOMES:
Particle size and distribution from exhaled breath | One year
  The exhaled air will be directed to a culturing media in place of the Sizer for collection of the droplets during two conditions: tidal breathing without oscillation (control) and tidal breathing with oscillation (experimental). The samples collected in the medium will later be cultured in a lab to determine the microbial species and their abundances. The purpose of Phase II experiments is to characterize the biological constituents produced from the oscillation enhanced sampling and contrast these constituents with those obtained during non-oscillation enhanced sampling. We hope to determine if the addition of oscillation increases the variety and abundance of microbial species able to be extracted from exhaled breath.

CONTACTS AND LOCATIONS:
Overall Officials: Erin P Silverman, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Afshar-Mohajer N, Wu CY, Tsai HW, Silverman E, Davenport P, Hegde S. Optimizing an Internal Airway Percussion Device for Facilitating Exhalate Diagnostics of the Human Respiratory System. J Aerosol Med Pulm Drug Deliv. 2015 Mar 31. [Epub ahead of print] PubMed PMID: 25826647.